CLINICAL TRIAL: NCT02189343
Title: A Phase 1b Multi-Center, Open Label, Dose-Escalation Study to Determine the Maximum Tolerated Dose, Safety, and Anti-Tumor Activity of an Alternative Liquid Formulation of ACY-1215 (Ricolinostat) In Combination With Pomalidomide and Low-Dose Dexamethasone In Patients With Relapsed and Refractory Multiple Myeloma
Brief Title: Phase 1b Study Evaluating ACY-1215 (Ricolinostat) in Combination With Pomalidomide and Dexamethasone in Relapsed or Relapsed-and-Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACE-MM-104
Record Dates: First submitted 2014-05-30; First posted 2014-07-14 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed and Refractory; Refractory Disease; Progressive Disease; Pomalidomide; Dexamethasone; Proteasome Inhibitor; Ricolinostat
MeSH Terms: conditions — Multiple Myeloma; Recurrence; Disease; Disease Progression | interventions — ricolinostat; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation Cohort (Experimental): Dose Escalating Cohorts of ACY-1215 in combination with pomalidomide and dexamethasone.
  Interventions: Drug: ACY-1215 in combination with pomalidomide and dexamethasone

INTERVENTIONS:
Drug: ACY-1215 in combination with pomalidomide and dexamethasone — Escalating dose Cohorts to determine a potential Maximum Tolerated Dose to recommend for a dosing schedule.
  Other Names: ACY-1215 (Ricolinostat); Pomalidomide; Dexamethasone

SUMMARY:
To determine the maximum tolerated dose (MTD), if present, and dose schedule of ACY-1215 (ricolinostat) in combination with pomalidomide and low-dose dexamethasone in patients with relapsed-and-refractory multiple myeloma.

DETAILED DESCRIPTION:
To determine the maximum tolerated dose (MTD), if present, and to identify a recommended dose and schedule of ricolinostat administered in an alternative liquid formulation (ALF) (10mg/mL) in combination with pomalidomide and low-dose dexamethasone in patients with relapsed or relapsed-and-refractory multiple myeloma.

To evaluate the safety and any anti-tumor activity of ricolinostat administered in combination with pomalidomide and dexamethasone as treatment for patients with relapsed or relapsed-and-refractory multiple myeloma, including duration of response.

To assess the Pharmacokinetics and Pharmacodynamics of all three medications administered in combination, and to assess the Pharmacokinetics of ricolinostat and pomalidomide specifically. An evaluation of the relationship between response and biomarkers relating to interacellular acetylation may also be completed.

ELIGIBILITY:
Key Inclusion Criteria Includes:

Patients meeting all of the following criteria may be enrolled in the study:

1. Must be able to understand and voluntarily sign an ICF.
2. Must be registered into the mandatory POMALYST Risk Evaluation and Mitigation Strategy (REMS)™ program, and be willing and able to comply with the requirements of the POMALYST REMS™ program (Appendix 9.3).
3. Must be ≥ 18 years of age at the time of signing the ICF.
4. Must be able to adhere to the study visit schedule and other protocol requirements.
5. Must have a documented diagnosis of MM and have relapsed or relapsed and refractory disease. Patients must have received at least 2 lines of prior therapies. Patients must have relapsed after having achieved at least stable disease for at least 1 cycle of treatment to at least 1 prior regimen and then developed PD. Relapsed and relapsed-and-refractory patients must have documented evidence of PD during or within 60 days (measured from the end of the last cycle) of completing treatment with the last antimyeloma drug regimen used just prior to study entry.
6. Patients must have undergone prior treatment with at least 2 cycles of lenalidomide and at least 2 cycles of a proteasome inhibitor (either in a separate regimen or within the same regimen.
7. Must not be a candidate for autologous stem cell transplant (ASCT), have declined the option of ASCT, or have relapsed after prior ASCT.
8. Must have measurable levels of myeloma paraprotein in serum (≥ 0.5 g/dL) or urine (≥ 0.2 g/24 hours). Patients who do not have myeloma paraprotein must have serum free light chain (SFLC) concentration of ≥ 10 mg/dL, provided SFLC ratio is abnormal. Nonsecretory myeloma is excluded.
9. Must have Eastern Cooperative Oncology Group performance status score of 0, 1, or 2.
10. Females of childbearing potential must have a negative serum or urine pregnancy test as described in Appendix 9.3 for the POMALYST REMS™ program. Females of childbearing potential and males must either commit to continued abstinence from heterosexual intercourse or must abide by birth control requirements as described in Appendix 9.3 for the POMALYST REMS™ program.
11. Must agree to refrain from donating blood while on study drug and for 28 days after discontinuation from this study.
12. Must agree not to share study medication with another person.
13. Must be able to take ASA (81 or 325 mg) daily as prophylactic anticoagulation. Patients intolerant to ASA may use low molecular weight heparin. Lovenox is recommended. Coumadin will be allowed provided the patient is fully anticoagulated, with an international normalized ratio of 2 to 3.

Key Exclusion Criteria Includes:

Patients meeting any of the following criteria will be excluded from enrollment in the study:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the ICF or from following the study requirements.
2. Pregnant or lactating females.
3. Prior therapy with histone deacetylase inhibitor or pomalidomide.
4. Any of the following laboratory abnormalities:

   * ANC < 1,000/µL
   * Platelet count < 75,000/ µL for patients in whom < 50% of bone marrow nucleated cells are plasma cells, or a platelet count < 50,000 for patients in whom ≥ 50% of bone marrow nucleated cells are plasma cells
   * Hemoglobin < 8 g/dL (< 4.9 mmol/L; prior red blood cell transfusion or recombinant human erythropoietin use is permitted).
   * Creatinine clearance < 45 mL/min according to Cockcroft-Gault formula. If creatinine clearance calculated from the 24 hour urine sample is ≥ 45 mL/min, patient will qualify for the trial.
   * Serum glutamic oxaloacetic transaminase/aspartate aminotransferase, or serum glutamic pyruvic transaminase/alanine aminotransferase > 3.0 × ULN
   * Serum total bilirubin > 2.0 mg/dL
5. Prior history of malignancies, other than MM, unless the patient has been free of the disease for ≥ 3 years. Exceptions include the following:

   * Basal or squamous cell carcinoma of the skin
   * Ductal carcinoma in situ; or cervical intraepithelial neoplasia
   * Carcinoma of the prostate with a current prostate-specific antigen below the upper limit of normal
6. Corrected QT interval (QTc) using Fridericia's formula value > 480 msec at Screening; family or personal history of long QTc syndrome or ventricular arrhythmias including ventricular bigeminy at Screening; previous history of drug-induced QTc prolongation or the need for treatment with medications known or suspected of producing prolonged QTc intervals on electrocardiogram.
7. Known human immunodeficiency virus, hepatitis B virus, and known or suspected active hepatitis C virus infection.
8. Hypersensitivity to thalidomide, lenalidomide, pomalidomide, or dexamethasone (such as Steven Johnson Syndrome). Hypersensitivity, such as rash, that can be medically managed is allowable.
9. Peripheral neuropathy ≥ Grade 2 despite supportive therapy.
10. Radiotherapy or systemic therapy (standard or an investigational or biologic anticancer agent) within 14 days of initiation of study drug treatment.
11. Current enrollment in another clinical trial involving treatment and/or receiving an investigational agent for any reason.
12. Inability or unwillingness to comply with birth control requirements or any of the POMALYST REMS™ requirements per Appendix 9.3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Determine Maximum Tolerated Dose (MTD) if any, and recommended dose schedule | Every 56 days on treatment, estimated average of 4 months.
  Identify the MTD of ACY-1215 administered in an alternative liquid formulation (ALF) if present, and identify a recommended dose and schedule. Patients will be followed for completion of 6 28-day Cycles of Study Treatment (for ITT Population analysis).

SECONDARY OUTCOMES:
Safety | Upon completion of a 28-day treatment cycle and for the duration of treatment, an estimated average of 4 months.
  To assess the type, frequency, and severity of adverse events (AEs) and relationship of AEs to study drug.
Anti-Tumor Activity | Upon completion of a 28-day treatment cycle and for the duration of treatment, an estimated average of 4 months.
  Anti-tumor activity will be measured by objective response to treatment as assessed by the site Investigators using International Myeloma Working Group (IMWG) Uniform Response criteria. Anti-tumor activity will also be measured by duration of response, time to response, and time to progression. The Response rate will be the percentage of patients who achieve PR or better. The number of patients who have at least MR or better will also be collected as clinical benefit response. Progression-free survival (PFS) will be defined as the time from first dose of study treatment to the first documentation of disease progression or death from any cause during the study. For responders, time to tumor response and response duration will be analyzed.
Pharmacokinetics | Up to 8 days post first dose
  Plasma levels of ACY-1215 will be measured to assess the single and multiple dose PK of AC-1215 in combination with pomalidomide and low-dose dexamethasone. Plasma levels of pomalidomide will be measured to assess the PK of pomalidomide in combination with ACY-1215 and low-dose dexamethasone.
Pharmacodynamics | Up to 24 hours post first dose
  Exposure response of ACY-1215 in combination with pomalidomide and low-dose dexamethasone, including biomarkers relating to intracellular protein acetylation, protein levels, mRNA and microRA expression profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Madan, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (3):
- United States (3):
  - UT Southwestern Medical Center Simmons Comprehensive Cancer Center, Dallas, Texas
  - CTRC at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah